CLINICAL TRIAL: NCT04708730
Title: Improving Neuroprotective Strategy for Ischemic Stroke After Thrombectomy Followed by DELP (INSIST-DELP): a Prospective, Random, Open-label, Blind-endpoint, Multi-centre Study
Brief Title: Improving Neuroprotective Strategy for Ischemic Stroke After Thrombectomy Followed by DELP (INSIST-DELP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Head of Neurology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y (2020) 043
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DELP (Experimental): Delipid Extracorporeal Lipoprotein filter from Plasma (DELP) is a non-pharmacological therapy for acute stroke, which is approved by China Food and Drug Administration
  Interventions: Device: Delipid Extracorporeal Lipoprotein filter from Plasma
- control group (No Intervention)

INTERVENTIONS:
Device: Delipid Extracorporeal Lipoprotein filter from Plasma — As a non-pharmacological therapy, Delipid Extracorporeal Lipoprotein filter from Plasma (DELP) hase been approved by China Food and Drug Administration to treat acute stroke
  Arms: DELP

SUMMARY:
Delipid Extracorporeal Lipoprotein filter from Plasma (DELP) has been found to improve neurological function and life ability of AIS patients and approved for the treatment of AIS by China Food and Drug Administration (CFDA). Our recent study imply that the neuroprotective effect of DELP involved multiple neuroprotective mechanism such as anti-inflammation, free radical scavenging, and decreasing MMP-9. Based on the multiple mechanisms, DELP was used to investigate the effect on acute ischemic stroke receiving endovascular treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* acute anterior circulatory cerebral infarction with large vessel occlusion;
* NIHSS≥6 before endovascular treatment;
* good recanalization (TICI 2b-3);
* time from onset to groin puncture is less than 8 hours;
* time from recanalization to DELP is less than 2 hours;
* Premorbid mRS 0 or 1;
* Signed informed consent.

Exclusion Criteria:

* poor recanalization (TICI 1-2a);
* Coagulation disorders, systematic hemorrhagic tendency, thrombocytopenia （ <100000/mm3;
* Severe hepatic or renal dysfunction, increase in ALT or AST (more than 2 times of upper limit of normal value), increase in serum creatinine (more than 1.5 times of upper limit of normal value) or requiring dialysis;
* Severe hypertension (systolic blood pressure over 200mmHg or diastolic blood pressure over 110 mmHg);
* Previous allergy to heparin or calcium;
* hypoproteinemia;
* Unsuitable for this clinical studies assessed by researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with modified Rankin Score 0 to 2 | Day 90

SECONDARY OUTCOMES:
Proportion of patients with modified Rankin Score 0 to 1 | Day 90
Changes in national institutes of health stroke scale (NIHSS) | 48 hours
  NIHSS ranges from 0-42, and the decrease in NIHSS means the improvement of neurological deficit.
Changes in national institutes of health stroke scale (NIHSS) | 7 days
  NIHSS ranges from 0-42, and the decrease in NIHSS means the improvement of neurological deficit.
Changes in cerebral infarct volume | 48 hours
the occurence of stroke or other cardiovascular events | Day 90
the occurence of infections post stroke | Day 14
Proportion of symptomatic intracranial hemorrhage (sICH) | 48 hours
  sICH was defined as 4 or more increase in NIHSS caused by hemorrhage
Proportion of intraparenchymal hemorrhage (PH1 and PH2) | 48 hours
the occurence of death due to any cause | Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared in request after the trial finish and will include study protocol, statistical analysis plan.
Supporting Information: Study Protocol, SAP, ICF, CSR